CLINICAL TRIAL: NCT05200000
Title: Evaluation of Wharton's Jelly Extract Eye Drops, Treated by the AMTRIX Process, in the Treatment of Chronic Keratitis
Brief Title: Wharton's Jelly Eye Drops in the Treatment of Chronic Keratitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SygeLIX-C-TBF1; 2019-A00866-51 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Keratitis, Ulcerative; Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SygeLIX-Coll-T (Experimental): Extract of umbilical cord lining constituted of Wharton's jelly put in suspension in microvials. Instillation by the patient in the sick eye of 1 drop 5 times a days (morning, noon, afternoon, evening and bedtime) for 40 days.
  Interventions: Biological: SygeLIX-Coll-T

INTERVENTIONS:
Biological: SygeLIX-Coll-T — Reconstituted suspension made of Trehalose and chemically treated, grinded, freeze-dried and sterilized Wharton's Jelly used by the patient as eye drops.

SUMMARY:
The purpose of this open, non-comparative, multicenter trial is to assess the impact of eye drops made of Wharton's jelly extract in the treatment of chronic keratitis that failed available therapies.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 70 years old.
* Persistent corneal ulceration.
* Resistance to medical treatment for more than one month or recurrence after medical treatment.
* Patient who underwent a wash-out period of 15 days with no use of eye drops with preservative.
* Patient with dry eye treatments that can be kept: tear substitutes, cyclosporine.
* Informed and consenting patient.
* Patient affiliated to a social security system or beneficiary of such a system.

Exclusion Criteria:

* Patient with active infectious or traumatic keratitis such as burns.
* Patient with herpetic keratitis.
* Patient currently wearing contact lens, including scleral lenses concomitant with the treatment.
* Patient currently treated with NSAIDs in eye drops or any eye drops containing preservatives.
* Patient treated with antibiotic, anti-viral or anti-parasitic eye drops; with autologous or allogeneic serum; with platelet derivatives; with eye drops claiming healing properties; with eye drops containing growth factors, hyaluronic acid or trehalose.
* Patient with hypersensitivity to fluorescein.
* Patient with identified causes for keratitis for which discontinuation of medical treatment is beneficial.
* Monophthalmic patients.
* Persons deprived of liberty by a judicial or administrative decision.
* Adults who are subject to a legal protection measure or who are unable to express their consent.
* Pregnant woman.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Absence of aggravated inflammatory signs, worsening of visual acuity or other side effect | Through study completion - average of 40 days
  Inflammatory signs evaluated using a composite score on 66 points. Duration and intensity are evaluated for secretion, dry eyes, tearing, foreign body sensation, fluctuating vision, photophobia, burning sensation and lids edema. Duration is evaluated from a scale from 0: never to 4: all the time. Intensity is evaluated from a scale from 0: slight to 2: severe. Localization and intensity are evaluated for conjunctival edema, conjunctival redness and neovascularization. Localization is evaluated on a scale from 0: no reaction to 4: reaction present in the whole eye

SECONDARY OUTCOMES:
Re-epithelialization of the cornea | 7 days, 15 days, 40 days
  Epithelialization assessed by the Oxford score after fluorescein instillation in the eye (0: no corneal staining to 5: severe corneal staining)
Improvement of dry eyes signs and symptoms | 7 days, 15 days, 40 days
  Severity of dry eye evaluated using Ocular Surface Disease Index (OSDI) questionnaire
Improvement of visual acuity | 7 days, 15 days, 40 days
  Visual acuity evaluated on Monoyer chart

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hôpital Michallon, CHU de Grenoble, La Tronche
  - Hôpital Gui de Chauliac, CHU de Montpellier, Montpellier
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - Hôpital Charles-Nicolle, CHU de Rouen, Rouen
  - Hôpital Nord, CHU de Saint-Etienne, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No